CLINICAL TRIAL: NCT06613243
Title: Different Doses of Dexmedetomidine Combined With Esketamine for Analgesia in Women Undergoing Cesarean Delivery: a Pilot Randomized Trial
Brief Title: Different Doses of Dexmedetomidine Combined With Esketamine in Women Undergoing Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, MD, PHD, Professor and Chairman, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-468
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Cesarean Delivery; Esketamine; Neuropsychiatric Symptoms; Dexmedetomidine
Keywords: cesarean delivery; esketamine; neuropsychiatric symptoms; dexmedetomidine
MeSH Terms: interventions — Esketamine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, pilot trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Esketamine 0.2 mg/kg (Active Comparator): Esketamine 0.2 mg/kg is diluted in 20 ml normal saline and infused over 40 minutes after clamping the umbilical cord.
  Interventions: Drug: Esketamine 0.2 mg/kg
- Esketamine 0.2 mg/kg + dexmedetomidine 0.1 µg/kg (Experimental): A mixture of esketamine 0.2 mg/kg and dexmedetomidine 0.1 µg/kg is diluted in 20 ml normal saline and infused over 40 minutes after clamping the umbilical cord.
  Interventions: Drug: Esketamine 0.2 mg/kg + dexmedetomidine 0.1 µg/kg
- Esketamine 0.2 mg/kg + dexmedetomidine 0.15 µg/kg (Experimental): A mixture of esketamine 0.2 mg/kg and dexmedetomidine 0.15 µg/kg is diluted in 20 ml normal saline and infused over 40 minutes after clamping the umbilical cord.
  Interventions: Drug: Esketamine 0.2 mg/kg + dexmedetomidine 0.15 µg/kg
- Esketamine 0.2 mg/kg + dexmedetomidine 0.2 µg/kg (Experimental): A mixture of esketamine 0.2 mg/kg and dexmedetomidine 0.2 µg/kg is diluted in 20 ml normal saline and infused over 40 minutes after clamping the umbilical cord.
  Interventions: Drug: Esketamine 0.2 mg/kg + dexmedetomidine 0.2 µg/kg

INTERVENTIONS:
Drug: Esketamine 0.2 mg/kg — Esketamine 0.2 mg/kg is diluted in 20 ml normal saline and infused over 40 minutes after clamping the umbilical cord.
  Arms: Esketamine 0.2 mg/kg
Drug: Esketamine 0.2 mg/kg + dexmedetomidine 0.1 µg/kg — A mixture of esketamine 0.2 mg/kg and dexmedetomidine 0.1 µg/kg is diluted in 20 ml normal saline and infused over 40 minutes after clamping the umbilical cord.
  Arms: Esketamine 0.2 mg/kg + dexmedetomidine 0.1 µg/kg
Drug: Esketamine 0.2 mg/kg + dexmedetomidine 0.15 µg/kg — A mixture of esketamine 0.2 mg/kg and dexmedetomidine 0.15 µg/kg is diluted in 20 ml normal saline and infused over 40 minutes after clamping the umbilical cord.
  Arms: Esketamine 0.2 mg/kg + dexmedetomidine 0.15 µg/kg
Drug: Esketamine 0.2 mg/kg + dexmedetomidine 0.2 µg/kg — A mixture of esketamine 0.2 mg/kg and dexmedetomidine 0.2 µg/kg is diluted in 20 ml normal saline and infused over 40 minutes after clamping the umbilical cord.
  Arms: Esketamine 0.2 mg/kg + dexmedetomidine 0.2 µg/kg

SUMMARY:
Esketamine is a commonly used analgesic during cesarean delivery, but may produce transient neuropsychiatric symptoms. Dexmedetomidine has both sedative and analgesic effects. When used in combination with esketamine, dexmedetomidine can reduce esketamine related neuropsychiatric effects after general anesthesia. The investigator speculate that combining low-dose dexmedetomidine with esketamine may also reduce neuropsychiatric adverse effects of esketamine in women undergoing cesarean section. This pilot trial is designed to determine the minimum dose of dexmedetomidine that can effectively prevent neuropsychiatric side effects of antidepressive dose esketamine (0.2mg/kg) in women undergoing cesarean delivery.

DETAILED DESCRIPTION:
Esketamine is a commonly used anesthetic and analgesic drug during the perioperative period. Recent studies found that low-dose esketamine has rapid onset antidepressant effects and reduces postpartum depression when administered during cesarean delivery. However, even low-dose esketamine produces transient neuropsychiatric symptoms.

Dexmedetomidine is a high selective alpha2-adrenoceptor agonist and has both sedative and analgesic effects. When used in combination with esketamine, dexmedetomidine reduces esketamine related neuropsychiatric adverse reactions in patients undergoing general anesthesia.

The investigator speculate that combining low-dose dexmedetomidine with esketamine may also reduce neuropsychiatric adverse effects of esketamine in women undergoing cesarean delivery. The purpose of this pilot trial is to determine the minimum dose of dexmedetomidine that can effectively prevent neuropsychiatric side effects of antidepressve dose esketamine (0.2mg/kg) in women undergoing cesarean delivery.

ELIGIBILITY:
Inclusion criteria:

* Pregnant women aged ≥18 years.
* Scheduled for elective or emergency cesarean delivery under neuraxial anesthesia.

Exclusion criteria:

* A previous history of schizophrenia;
* Severe complications of pregnancy, such as pre-eclampsia, placenta accreta spectrum, or HELLP (intravascular haemolysis, elevated liver enzymes, and low platelet count) syndrome; or American Society of Anesthesiologists classification III or higher;
* Any contraindications to ketamine or esketamine, such as refractory hypertension, severe cardiovascular disease, or hyperthyroidism;
* Any contraindications to dexmedetomidine, such as sick sinus syndrome, severe sinus bradycardia (<50 beats per minute), or second-degree or above atrioventricular block without pacemaker;
* Other conditions that are considered unsuitable for study participation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Incidence of dissociation within 24 hours. | Up to 24 hours after study drug infusion.
  Dissociative symptoms is assessed with the Clinician-Administered Dissociative States Scale (CADSS; scores range from 0 to 92, with higher score indicating more severe symptoms) at the end of study drug infusion and at 1, 2, and 24 hours after study drug infusion. A CADSS score of >4 points at any timepoint indicates occurrence of dissociative symptoms.

SECONDARY OUTCOMES:
Severity of dissociative symptoms at different timepoints within 24 hours. | Up to 24 hours after study drug infusion.
  Dissociation symptoms is assessed with the Clinician-Administered Dissociative States Scale (CADSS; scores range from 0 to 92, with higher score indicating more severe symptoms) at the end of study drug infusion and at 1, 2, and 24 hours after study drug infusion.
Prevelance of dissociation at different timepoints within 24 hours. | Up to 24 hours after study drug infusion.
  Dissociation symptoms is assessed with the Clinician-Administered Dissociative States Scale (CADSS; scores range from 0 to 92, with higher score indicating more severe symptoms) at the end of study drug infusion and at 1, 2, and 24 hours after study drug infusion.
Incidence of neuropsychiatric adverse events within 24 hours. | Up to 24 hours after study drug infusion.
  Neuropsychiatric symptoms are evaluated with a structured checklist at 5-minute intervals during, at 10-minute intervals after, and at 2 and 24 hours after study drug infusion. Severity of symptoms is classified as mild (report symptoms on inquiry), moderate (report symptoms without inquiry), or severe (required intervention such as stop study drug infusion and/or give medications). A severity of moderate or above is recorded as presence of neuropsychiatric symptoms.
Prevalence of neuropsychiatric adverse events at different timepoints within 24 hours. | Up to 24 hours after study drug infusion.
  Neuropsychiatric symptoms are evaluated with a structured checklist every 5 minutes during, every 10 minutes after, and at 2 and 24 hours after study drug infusion. Severity of symptoms is classified as mild (report symptoms on inquiry), moderate (report symptoms without inquiry), or severe (required intervention such as stop study drug infusion and/or give medications). A severity of moderate or above is defined as presence of neuropsychiatric symptoms.

OTHER OUTCOMES:
Duration of sedation within 24 hours. | Up to 24 hours after study drug infusion.
  Agitation-sedation level is assessed with the Richmond Agitation-Sedation Scale (RASS, score ranges from -5 [unarousable] to 4 [combative] and 0 indicates alert and calm) and recorded every 5 minutes during, every 10 minutes after, and at 2 hours and 24 hours after study drug infusion. A RASS score of <-1 is defined as presence of sedation.
Pain intensity within 7 days postpartum. | Up 7 days postpartum.
  Pain intensity is assessed with the Numeric Rating Scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain), both at rest and with movement, at 2 and 24 hours after study drug infusion and at 7 days postpartum.
Proportion of exclusive breastfeeding. | Up to 7 days postpartum.
  Proportion of exclusive breastfeeding at 24 hours and 7 days postpartum.
Length of stay in hospital after surgery. | Up to 7 days postpartum.
  Length of stay in hospital after surgery.
Maternal and neonatal complications within 7 days. | Up to 7 days postpartum.
  Maternal and neonatal complications are defined as any medical conditions that required hospital visits and therapeutic intervention.
Maternal depression score at 7 days postpartum. | At 7 days postpartum.
  Maternal depression is assessed with the Edinburgh Postnatal Depression Scale (EPDS; scores range from 0 to 30, with higher score indicating more severe depression) at 7 days postpartum. An EPDS score of ≥10 is defined as having depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, M.D., PhD., Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bremner JD, Krystal JH, Putnam FW, Southwick SM, Marmar C, Charney DS, Mazure CM. Measurement of dissociative states with the Clinician-Administered Dissociative States Scale (CADSS). J Trauma Stress. 1998 Jan;11(1):125-36. doi: 10.1023/A:1024465317902. PMID 9479681
- [Background] Keating GM. Dexmedetomidine: A Review of Its Use for Sedation in the Intensive Care Setting. Drugs. 2015 Jul;75(10):1119-30. doi: 10.1007/s40265-015-0419-5. PMID 26063213
- [Background] Daly EJ, Singh JB, Fedgchin M, Cooper K, Lim P, Shelton RC, Thase ME, Winokur A, Van Nueten L, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine Adjunctive to Oral Antidepressant Therapy in Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):139-148. doi: 10.1001/jamapsychiatry.2017.3739. PMID 29282469
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Lu X, Tang L, Lan H, Li C, Lin H. A Comparison of Intranasal Dexmedetomidine, Esketamine or a Dexmedetomidine-Esketamine Combination for Induction of Anaesthesia in Children: A Randomized Controlled Double-Blind Trial. Front Pharmacol. 2022 Jan 27;12:808930. doi: 10.3389/fphar.2021.808930. eCollection 2021. PMID 35185548
- [Background] Mello RP, Echegaray MVF, Jesus-Nunes AP, Leal GC, Magnavita GM, Vieira F, Caliman-Fontes AT, Telles M, Guerreiro-Costa LNF, Souza-Marques B, Bandeira ID, Santos-Lima C, Marback RF, Correia-Melo FS, Lacerda ALT, Quarantini LC. Trait dissociation as a predictor of induced dissociation by ketamine or esketamine in treatment-resistant depression: Secondary analysis from a randomized controlled trial. J Psychiatr Res. 2021 Jun;138:576-583. doi: 10.1016/j.jpsychires.2021.05.014. Epub 2021 May 8. PMID 33991996
- [Background] Zhang Y, Cui F, Ma JH, Wang DX. Mini-dose esketamine-dexmedetomidine combination to supplement analgesia for patients after scoliosis correction surgery: a double-blind randomised trial. Br J Anaesth. 2023 Aug;131(2):385-396. doi: 10.1016/j.bja.2023.05.001. Epub 2023 Jun 9. PMID 37302963
- [Background] Wang S, Deng CM, Zeng Y, Chen XZ, Li AY, Feng SW, Xu LL, Chen L, Yuan HM, Hu H, Yang T, Han T, Zhang HY, Jiang M, Sun XY, Guo HN, Sessler DI, Wang DX. Efficacy of a single low dose of esketamine after childbirth for mothers with symptoms of prenatal depression: randomised clinical trial. BMJ. 2024 Apr 10;385:e078218. doi: 10.1136/bmj-2023-078218. PMID 38808490
- [Background] Yang JR, Li YY, Ran TJ, Lin XY, Xu JY, Zhou SL, Huang PJ. Esketamine Combined with Dexmedetomidine to reduce Visceral Pain During elective Cesarean Section Under Combined Spinal-Epidural Anesthesia: A double-Blind Randomized Controlled Study. Drug Des Devel Ther. 2024 Jun 18;18:2381-2392. doi: 10.2147/DDDT.S460924. eCollection 2024. PMID 38911034